CLINICAL TRIAL: NCT04191421
Title: A Phase Ib/II Trial of Siltuximab and Spartalizumab in Metastatic Pancreatic Cancer
Brief Title: Siltuximab and Spartalizumab in Patients With Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Novartis (Industry); EUSA Pharma, Inc. (Industry); National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Olatunji Alese, Principal Investigator, Emory University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB00105616; NCI-2018-01793 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Winship4463-18 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2019-12-05; First posted 2019-12-09 (Actual); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Pancreatic Adenocarcinoma; Stage IV Pancreatic Cancer AJCC v8
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — siltuximab; spartalizumab

STUDY DESIGN:
Intervention Model Description: Arm 1- (Phase I dose level 1)- Siltuximab 6 mg/Kg every 3 weeks and Spartalizumab 300mg every 3 weeks Arm 2- (Phase I dose level 2)- Siltuximab 11 mg/Kg every 3 weeks and spartalizumab 300 mg every 3weeks Arm 3 - (Phase I doe level 2a)- Siltuximab 9 mg/Kg every 3 weeks and spartalizumab 300 mg every 3weeks Arm 4- (Phase II)- Siltuximab RP2D determined in Arms 1 to 3 and spartalizumab 300 mg every 3weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment spartalizumab and siltuximab Phase I dose level 1 (Experimental): Arm 1 (Phase I dose level 1) Participants receive spartalizumab 300 mg IV over 30 minutes on day 1 and siltuximab 6 mg/Kg IV over 1 hour on day 1. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Siltuximab; Biological: Spartalizumab
- Treatment spartalizumab and siltuximab Phase I level 2 (Experimental): Arm 2 (Phase I dose level 2) Participants receive spartalizumab 300 mg IV over 30 minutes on day 1 and siltuximab 11 mg/Kg IV over 1 hour on day 1. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Siltuximab; Biological: Spartalizumab
- Treatment spartalizumab and siltuximab phase I level 2a (Experimental): Arm 3 (Phase I dose level 2a) Participants receive spartalizumab 300 mg IV over 30 minutes on day 1 and siltuximab 9 mg/Kg IV over 1 hour on day 1. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Siltuximab; Biological: Spartalizumab
- Treatment spartalizumab and siltuximab phase II (Experimental): Arm 4 (Phase II ) Participants receive spartalizumab 300 mg IV over 30 minutes on day 1 and siltuximab at dose determined in Arm 1 to 3 IV over 1 hour on day 1. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Siltuximab; Biological: Spartalizumab

INTERVENTIONS:
Biological: Siltuximab — Given IV
  Other Names: Anti-IL-6 Chimeric Monoclonal Antibody; cCLB8; CNTO 328; Sylvant
Biological: Spartalizumab — Given IV
  Other Names: PDR001

SUMMARY:
This phase Ib/II trial studies the best dose and side effects of siltuximab and how well it works in combination with spartalizumab in treating patients with pancreatic cancer that has spread to other places in the body. Monoclonal antibodies, such as siltuximab and spartalizumab, interfere with the ability of tumors cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the recommended phase II dose for the combination of spartalizumab and siltuximab.

SECONDARY OBJECTIVES:

I. Define the toxicity profile of the combination of the recommended phase II dose of spartalizumab and siltuximab.

II. Evaluate the activity of the combination of spartalizumab and siltuximab in previously treated patients with pancreatic cancer.

EXPLORATORY OBJECTIVE:

I. Evaluate the effect of the combination on the immune profile in the serum and in tumor biopsies.

OUTLINE: This is a dose-escalation study of siltuximab.

Participants receive spartalizumab intravenously (IV) over 30 minutes on day 1 and siltuximab IV over 1 hour on day 1. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up at 30, 60, 90, 120, and 150 days, then every 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Cytological or histologic diagnosis and metastatic pancreatic adenocarcinoma disease that has failed at least one standard regimen such as gemcitabine nab-paclitaxel or folinic acid, fluorouracil, irinotecan hydrochloride, and oxaliplatin (FOLFIRINOX).
* Patient must meet the following laboratory values at the screening visit:

  * Absolute neutrophil count ≥ 1.5 x 109/L
  * Platelets ≥ 75 x 109/L
  * Hemoglobin (Hgb) ≥ 9 g/dL
  * Serum creatinine < 1.5 mg/dL OR Creatinine Clearance ≥ 45 mL/min using Cockcroft-Gault formula
  * Total bilirubin ≤ 1.5 x ULN
  * Aspartate transaminase (AST) ≤ 2.5 x ULN, except for patients with liver metastasis, who may only be included if AST ≤ 5.0 x upper limit of normal (ULN)
  * Alanine transaminase (ALT) ≤ 2.5 x ULN, except for patients with liver metastasis, who may only be included if ALT ≤ 5.0 x ULN
* Presence of measurable disease by RECIST criteria
* Patient has an Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Written informed consent must be obtained prior to any screening procedures.
* Normal ECG defined as the following:
* Resting heart rate 50-90 bpm
* QT corrected for HR using Fridericia's method (QTcF) at screening < 450 ms (male patients), < 460 ms (female patients)
* Before enrollment, a woman must be either:

  * Not of childbearing potential: postmenopausal (> 45 years of age with amenorrhea for at least 12 months or any age with amenorrhea for at least 6 months and a serum follicle stimulating hormone (FSH) level > 40 IU/mL); permanently sterilized (eg, tubal occlusion, hysterectomy, bilateral salpingectomy); or otherwise be incapable of pregnancy
  * Of childbearing potential and practicing (during the study and for 150 days after receiving the last dose of study agent) a highly effective method of birth control consistent with local regulations regarding the use of birth control methods for subjects participating in clinical studies: eg, established use of oral, injected or implanted hormonal methods of contraception; placement of an intrauterine device (IUD) or intrauterine system (IUS); barrier methods: condom with spermicidal foam/gel/film/cream/suppository or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository; male partner sterilization (the vasectomized partner should be the sole partner for that subject); true abstinence (when this is in line with the preferred and usual lifestyle of the subject)
  * Note: If the childbearing potential changes after start of the study (eg, woman who is not heterosexually active becomes active) a woman must begin a highly effective method of birth control, as described above.
* A woman of childbearing potential must have a negative serum (β-human chorionic gonadotropin [β-hCG]) or urine pregnancy test at screening.
* During the study and for 150 days after receiving the last dose of study agent, a woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction.
* A man who is sexually active with a woman of childbearing potential and has not had a vasectomy must agree to use a barrier method of birth control eg, either condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository, and all men must also not donate sperm during the study and for 3 months after receiving the last dose of study drug.
* Sign an informed consent document indicating that they understand the purpose of and procedures required for the study, are willing to participate in the study, and are willing and able to adhere to the prohibitions and restrictions specified in this protocol. Informed consent must be obtained before performing any study specific procedures.

Exclusion Criteria:

* Prior exposure to agents targeting programmed cell death protein-1 (PD-1), PD-L1, IL-6 or the IL-6 receptor. Prior chemotherapy is allowed as long as adequate washout period of ≥ 4 weeks.
* Any untreated central nervous system (CNS) lesion. However, patients are eligible if: a) all known CNS lesions have been treated with radiotherapy or surgery and b) patient remained without evidence of CNS disease progression ≥ 4 weeks after treatment and c) patients must be off corticosteroid therapy for ≥ 2 weeks.
* Use of any live vaccines against infectious diseases within 4 weeks of initiation of study treatment.
* Systemic chronic steroid therapy (≥ 10mg/day prednisone or equivalent) or any immunosuppressive therapy 7 days prior to planned date of first dose of study treatment. Note: Topical, inhaled, nasal and ophthalmic steroids are allowed.
* Active, known or suspected autoimmune disease or a documented history of autoimmune disease Note: Patients with vitiligo, controlled type I diabetes mellitus on stable insulin dose, residual autoimmune-related hypothyroidism only requiring hormone replacement or psoriasis not requiring systemic treatment are permitted).
* Allogenic bone marrow or solid organ transplant.
* History of severe hypersensitivity reactions to other monoclonal antibodies, which in the opinion of the investigator may pose an increased risk of serious infusion reaction.
* Known history or current interstitial lung disease or non-infectious pneumonitis.
* Malignant disease, other than that being treated in this study. Exceptions to this exclusion include the following: malignancies that were treated curatively and have not recurred within 2 years prior to study treatment; completely resected basal cell and squamous cell skin cancers and any completely resected carcinoma in situ.
* Clinically significant infection, including known HIV or hepatitis C infection, or known hepatitis B surface antigen positivity.
* Clinically significant ongoing infection.
* Received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 14 days or 5 half-lives before enrollment (whichever is longer) or is currently enrolled in the treatment stage of an investigational study.
* A woman who is pregnant or breast-feeding, or a woman who is planning to become pregnant or a man who plans to father a child while enrolled in this study or within 150 days after the last dose of study agent.
* Had hospitalization for infection or major surgery (eg, requiring general anesthesia) within 2 weeks before enrollment or have not fully recovered from surgery. Note: subjects with surgical procedures conducted under local anesthesia may participate.
* History or current diagnosis of cardiac disease indicating significant risk of safety for patients participating in the study such as uncontrolled or significant cardiac disease, including any of the following:

  * Recent myocardial infarction (within last 6 months)
  * Uncontrolled congestive heart failure
  * Unstable angina (within last 6 months)
  * Clinically significant (symptomatic) cardiac arrhythmias (e.g., sustained ventricular tachycardia, and clinically significant second or third degree atrioventricular block (AV) block without a pacemaker)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2023-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olatunji Alese, MD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Treatment Spartalizumab and Siltuximab Phase I Level 2: Arm 2 (Phase I dose level 2) Participants receive spartalizumab 300 mg IV over 30 minutes on day 1 and siltuximab 11 mg/Kg IV over 1 hour on day 1. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Siltuximab: Given IV
  Spartalizumab: Given IV
Period: Overall Study
Arm/Group | Treatment Spartalizumab and Siltuximab Phase I Dose Level 1 | Experimental: Treatment Spartalizumab and Siltuximab Phase I Level 2
Started | 4 | 31
Completed | 4 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Spartalizumab and Siltuximab RP2D: Arm 2 (Phase I dose level 2) Participants receive spartalizumab 300 mg IV over 30 minutes on day 1 and siltuximab 11 mg/Kg IV over 1 hour on day 1. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Siltuximab: Given IV
  Spartalizumab: Given IV
- Total: Total of all reporting groups
Arm/Group | Treatment Spartalizumab and Siltuximab Phase I Dose Level 1 | Treatment Spartalizumab and Siltuximab RP2D | Total
Number analyzed (Participants) | 4 | 31 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 12 | 14
  >=65 years | 2 | 19 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 17 | 20
  Male | 1 | 14 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 25 | 29
  Unknown or Not Reported | 0 | 6 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 1 | 22 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 4 | 31 | 35

OUTCOME MEASURES:

1. Primary Outcome: Maximal Tolerated Dose (MTD) of Siltuximab That Can be Combined With Spartalizumab
Description: Maximal tolerated dose (MTD )is defined as the dose at which less than one-third of the subjects experience a dose-limiting toxicity (DLT) in the first 6 weeks of treatment. A DLT is defined as an adverse event or abnormal laboratory value assessed as definitely at least possibly related to study treatment treatment related that occurs within the first 6 weeks. National Cancer Institute Common Terminology Criteria for Adverse events (NCI CTCAE) version 4.03 will be used for all grading.
Time Frame: Up to 6 weeks from study start
Measure: Number; unit: mg/kg
Arm/Group | Treatment Spartalizumab and Siltuximab Phase I Dose Level 1
Number analyzed (Participants) | 35
mg/kg | 11

2. Secondary Outcome: Overall Response Rate (ORR)
Description: Overall response rate is defined as complete response (CR) + partial response (PR) in participants treated with siltuximab and spartalizumab and will be assessed by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
Time Frame: Up to 2 years from study start
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment Spartalizumab and Siltuximab Phase I Dose Level 1 | Treatment Spartalizumab and Siltuximab RP2D
Number analyzed (Participants) | 4 | 31
percentage of participants | 0 [0 to 0] | 0 [0 to 0]

3. Secondary Outcome: Response Duration
Description: Will be assessed by RECIST 1.1.
Time Frame: From treatment start until progression or death, assessed up to 2 years
Population: No patients achieved CR/PR. The response duration cannot be evaluated.
Groups:
- Treatment Spartalizumab and Siltuximab: Arm 1 (Phase I dose level 1) Participants receive spartalizumab 300 mg IV over 30 minutes on day 1 and siltuximab 6 mg/Kg IV over 1 hour on day 1. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Siltuximab: Given IV
  Spartalizumab: Given IV
Arm/Group | Treatment Spartalizumab and Siltuximab | Treatment Spartalizumab and Siltuximab RP2D
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Progression-free Survival
Description: Will be assessed by RECIST 1.1.
Time Frame: From treatment start until progression or death, assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment Spartalizumab and Siltuximab Phase I Dose Level 1 | Treatment Spartalizumab and Siltuximab RP2D
Number analyzed (Participants) | 4 | 31
months | 1.9 [1.6 to NA] — Upper CI was non-evaluable due to insufficient participants with events for DL-1. | 2.1 [1.5 to 2.2]

5. Secondary Outcome: Overall Survival Time
Description: Will be assessed by RECIST 1.1.
Time Frame: From treatment start until progression or death, assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment Spartalizumab and Siltuximab Phase I Dose Level 1 | Treatment Spartalizumab and Siltuximab RP2D
Number analyzed (Participants) | 4 | 31
months | 9.3 [5.3 to NA] — Upper CI was non-evaluable due to insufficient participants with events for DL-1. | 3.1 [1.9 to 5.6]

ADVERSE EVENTS:
Time Frame: 24 months
Groups:
- Treatment Spartalizumab and Siltuximab Phase I Dose Level 1: Arm 1 (Phase I dose level 1) Participants receive spartalizumab 300 mg IV over 30 minutes on day 1 and siltuximab 6 mg/Kg IV over 1 hour on day 1. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Siltuximab: Given IV Spartalizumab: Given IV
Arm/Group | Treatment Spartalizumab and Siltuximab Phase I Dose Level 1 | Experimental: Treatment Spartalizumab and Siltuximab Phase I Level 2
All-Cause Mortality (participants affected / at risk) | 4/4 | 26/31
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/31
Other Adverse Events (participants affected / at risk) | 2/4 | 15/31
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Spartalizumab and Siltuximab Phase I Dose Level 1 (N=4) | Experimental: Treatment Spartalizumab and Siltuximab Phase I Level 2 (N=31)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhea (Investigations) | 0 (0) | 1 (1)
Flatulence (Nervous system disorders) | 0 (0) | 1 (1)
Vomiting (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Fatigue (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
General Disorders-other (General disorders) | 0 (0) | 2 (2)
Hepatic Failure (General disorders) | 0 (0) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 3 (3)
Alanine aminotransferase increased (General disorders) | 0 (0) | 3 (3)
Alkaline phosphatase increased (General disorders) | 0 (0) | 3 (3)
Blood Bilirubin Increased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (General disorders) | 0 (0) | 1 (1)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-15): https://cdn.clinicaltrials.gov/large-docs/21/NCT04191421/Prot_SAP_002.pdf
  • Informed Consent Form (2023-01-20): https://cdn.clinicaltrials.gov/large-docs/21/NCT04191421/ICF_003.pdf